CLINICAL TRIAL: NCT04222855
Title: Efficacy of Diltiazem for the Control of Blood Pressure in Puerperal Patients With Severe Preeclampsia: A Randomized Controlled Trial
Brief Title: Efficacy of Diltiazem for the Control of Blood Pressure in Puerperal Patients With Severe Preeclampsia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de la Mujer (Other Government)
Collaborators: Ocharan-Hernández, Esther, MD, PhD (Unknown); Vargas-De-León, Cruz, MSc (Unknown); Calzada-Mendoza, Claudia, PhD (Unknown)
Responsible Party: Principal Investigator, Dr. Gilberto Arias-Hernández, Physician of the Intensive Care Unit, Hospital de la Mujer
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CCINSHAE-DGCHFR-HMD-DEI-2008
Record Dates: First submitted 2020-01-07; First posted 2020-01-10 (Actual); Last update posted 2020-01-10 (Actual); Status verified 2020-01

CONDITIONS: Postpartum Preeclampsia
MeSH Terms: interventions — Diltiazem

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diltiazem (Experimental): Postpartum patients were administered (60 mg) orally every 8 hours with diltiazem (tables).
  Interventions: Drug: Diltiazem
- Nifedipine (Active Comparator): Postpartum patients were administered (10 mg) orally every 8 hours with nifedipine (capsule).
  Interventions: Drug: Diltiazem

INTERVENTIONS:
Drug: Diltiazem — Puerperal patients was administered (60 mg) orally every 8 hours with diltiazem (tables).

SUMMARY:
Both preeclampsia and eclampsia are important health problems, being an important cause of maternal death in the world.

Nifedipine has been used as the drug of choice for the treatment of hypertension during puerperium for more than 25 years.

Diltiazem is an alternative calcium antagonist that is 1000 times less potent than nifedipine.

There are no reports in the literature, no randomized clinical trials that prove the effectiveness of diltiazem for the control of blood pressure in post-partum patients with severe preeclampsia.

DETAILED DESCRIPTION:
Both preeclampsia and eclampsia are important health problems, being an important cause of maternal death in the world. Although these two pregnancy-related disorders have been widely studied, their cause remains unknown. Pathophysiological mechanism involves the reduction of maternal placental blood flow as of week 20 of gestation, with an increase in peripheral vascular resistance that predominantly takes place in the kidney, liver and brain.

Nifedipine has been used as the drug of choice for the treatment of hypertension during puerperium for more than 25 years. However, there are various studies that report in sensible population the presence of serious adverse effects with the use of this drug, such as cerebral ischemia, myocardial ischemia or tachycardia, as well as episodes of hyper- and hypotension. Consequently, it is necessary to find treatment alternatives for this case.

Diltiazem is an alternative calcium antagonist that is 1000 times less potent than nifedipine, which has the property of producing a selective vasodilatation of arteries beds.

There are no reports in the literature, no randomized clinical trials that prove the effectiveness of diltiazem for the control of blood pressure in post-partum patients with severe preeclampsia.

The objective of this study is to evaluate if diltiazem improves the blood pressure parameters in early puerperium patients with severe preeclampsia.

A researcher who was not involved in the study was performed the randomization by using a random- numbers table and central allocation. All participants and study staff were blind to medication condition. The patients were randomly allocated to one of two groups of treatment: group one was administered 60 mg of diltiazem (tables) while group two (the control) was administered 10 mg of nifedipine (capsule). Both drugs were administered orally every 8 hours. Systolic, diastolic and mean blood pressures and heart rate were recorded and analyzed at baseline and 6, 12, 18, 24, 30, 36, 42 and 48 hours.

A Foley catheter was placed to measure urinary excretion. On the other hand, the blood pressure of all patients was continuously recorded using a monitor (DASH 4000 Dinamar, US) which provided a reading of systolic, diastolic and mean blood pressure trough central venous catheter. The register was taken during the 48-hour observation period, in order to ensure that blood pressure was maintained between 120/70 and 160/110 mmHg; either determine hypotension (which is defined by the pressure at which clinical alterations occur) or hypertension events.

The size of the sample was calculated with the formula of difference between the means of two independent samples. We took the systolic pressure values from a pilot study of 10 subjects for each group. The common standard deviation of delta values (Baseline and after 72-hour pressure difference) is 19 mmHg, a difference between delta values of the treatments is 16.5 mmHg, and a power level of 0.8, resulting in 21 patients per group.

Comparisons between groups on the repeated measures were made using repeated-measure ANOVA. Analyses included fixed effects for time (baseline and 6, 12, 18, 24, 30, 36, 42 and 48 hours) and treatments (diltiazem and nifedipine), and treatments×time interactions. If the interaction was statistically significant, post hoc analysis using the Sidak correction method for mean differences were used to determine whether the changes in levels of arterial blood pressure between the longitudinal assessments were statistically significant between the diltiazem and nifedipine treatments. When necessary, a Greenhouse-Geisser correction was applied to correct for non-sphericity.

ELIGIBILITY:
Inclusion Criteria:

The following parameters of all patients were within the normal range: hematic biometry, urine and glucose tests, aspartate aminotransferase (AST), alanine aminotransferase (ALT), serum creatinine, blood coagulation test including prothrombin time and activated partial thromboplastin time. Electrocardiogram and chest radiography showed no pathological data.

Exclusion Criteria:

When the patient falls outside of the aforementioned parameters, or subjects with unstable medical conditions.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2009-01-01 (Actual); Primary Completion 2009-05-30 (Actual); Study Completion 2009-05-30 (Actual)

PRIMARY OUTCOMES:
Systolic blood pressure | The register was taken during the 48-hour observation period
Diastolic blood pressure | The register was taken during the 48-hour observation period
Mean blood pressure | The register was taken during the 48-hour observation period

SECONDARY OUTCOMES:
Number of hypotension episodes | The counts was taken during the 48-hour observation period
Days of stay in the intensive care unit | The counts was taken during the two-weeks observation period

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Arias-Hernandez G, Vargas-De-Leon C, Calzada-Mendoza CC, Ocharan-Hernandez ME. Efficacy of Diltiazem for the Control of Blood Pressure in Puerperal Patients with Severe Preeclampsia: A Randomized, Single-Blind, Controlled Trial. Int J Hypertens. 2020 Jul 23;2020:5347918. doi: 10.1155/2020/5347918. eCollection 2020. PMID 32774912